CLINICAL TRIAL: NCT05499221
Title: Segmental Distalization by Bone Anchored Carriere Motion Appliance vs. Conventional One
Brief Title: Bone Anchored Carriere Motion Appliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eglal Ahmed, Dr., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A01040122
Record Dates: First submitted 2022-08-05; First posted 2022-08-12 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Malocclusion, Angle Class II
Keywords: Carriere motion appliance; Distalization; Skeletal anchorage; Infrazygomatic miniscrews
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated into two groups:
  1. Conventional anchorage CMA group (CAG): conventional mandibular anchorage using Essix retainer.
  2. Skeletal anchorage CMA group (SAG): anchorage by infra-zygomatic mini-screws. In the CAG, Class II elastics will be attached from the maxillary canine to the mandibular first molar bilaterally with Essix retainer in the lower arch as anchorage means. In the SAG, the closing coil spring will be attached from the maxillary canine to the infra zygomatic miniscrews bilaterally. For each patient, two lateral cephalograms will be obtained: one preoperatively and another after completion of distalization. Model measurements will be made using the attached 3Shape computer software.
Who Masked: Outcomes Assessor
Masking Description: data will be sent blinded for statistical analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional anchorage (Active Comparator): Buccal tubes will be bonded on the lower first molars, an alginate impression will be taken for the lower arch with the buccal tubes in place, and a cast will be poured. A hard vacuum sheet of 1.5- mm thickness will be used to fabricate the Essix appliance. The posterior end of the buccal surface will be trimmed in each lower first molar region, creating a window to allow for attachment of the elastics. Class II elastics will be attached from the maxillary canine to the mandibular first molar bilaterally. During the first month, 1/4-inch heavy elastics will be used. In the following months, 3/16-inch heavy elastics will be used. The patients will be instructed to wear the elastics 24 hours per day, except during mealtimes, and to change them daily.
  Interventions: Device: Carriere motion appliance
- Skeletal anchorage (Experimental): Closing coil springs will be attached from the maxillary canine to the infrazygomatic miniscrews bilaterally
  Interventions: Device: Carriere motion appliance

INTERVENTIONS:
Device: Carriere motion appliance — The CMA will be bonded on the permanent maxillary canine and first molar, and the correct size is chosen according to the manufacturer's instructions.

SUMMARY:
Carriere Motion appliance (CMA) was designed to change a Class II molar relationship into a Class I relationship by distalizing the whole posterior maxillary segment by means of class II elastics and mandibular anchorage. To eliminate the adverse effects of CMA with class II elastics, we can use the CMA to distalize the maxillary posterior segment with intra-arch anchorage using infrazygomatic miniscrews. The aim of this study is to evaluate skeletaly anchored CMA for distalization of the maxillary buccal segment vs. conventionally anchored CMA by comparing skeletal and dental measurements obtained from lateral cephalometric radiographs obtained prior to treatment (T0) and immediately after correction of class II and remval of the appliance (T1).

DETAILED DESCRIPTION:
Thirty-two class II malocclusion patients with age (11-16) years will be randomly allocated in the two groups:

1. Conventional anchorage CMA group (CAG): conventional mandibular anchorage using Essix retainer.
2. Skeletal anchorage CMA group (SAG): anchorage by infra-zygomatic miniscrews. In the CAG, Class II elastics will be attached from the maxillary canine to the mandibular first molar bilaterally with Essix retainer in the lower arch as anchorage means. In the SAG, closing coil spring will be attached from the maxillary canine to the infrazygomatic miniscrews bilaterally. For each patient, two lateral cephalograms will be obtained: one preoperatively and another after completion of distalization. Model measurements will be made using the attached 3Shape computer software.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age (11-16) years.
2. Full permanent dentition.
3. Class II malocclusion with at least an end-on Class II molar relationship bilaterally.

Exclusion Criteria:

1. Systemic conditions that may interfere with the treatment.
2. Bad habits that might jeopardize the appliance.
3. Transverse discrepancy.
4. Previous orthodontic treatment.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Treatment duration | from date of appliance delivery to date of removal after reaching class I molar relationship (about 4-6 months)
  months
Skeletal changes | from date of appliance delivery to date of removal after reaching class I molar relationship (about 4-6 months)
  degrees
Dental changes | from date of appliance delivery to date of removal after reaching class I molar relationship (about 4-6 months)
  degrees

CONTACTS AND LOCATIONS:
Overall Officials: Eglal A. Ghozy, BDS, MDS, Principal Investigator — Mansoura University; Ahmed A. El-bialy, PhD, Study Chair — Mansoura University; Marwa S. Shamaa, PhD, Study Director — Mansoura University; Nehal F. Albelasy, PhD, Study Director — Mansoura University
Locations (1):
- MansouraU, faculty of dentistry, orthodontics department, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghozy EA, Albelasy NF, Shamaa MS, El-Bialy AA. Cephalometric and digital model analysis of dentoskeletal effects of infrazygomatic miniscrew vs. Essix- anchored Carriere Motion appliance for distalization of maxillary buccal segment: a randomized clinical trial. BMC Oral Health. 2024 Jan 31;24(1):152. doi: 10.1186/s12903-024-03925-3. PMID 38297285